CLINICAL TRIAL: NCT05489575
Title: Hemodynamic Effects of Positive Airway Pressure to Treat Supine Hypertension and Improve Neurogenic Orthostatic Hypotension
Brief Title: CPAP for the Treatment of Supine Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor of Medicine and Pharmacology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 220821; R01HL161095 (NIH); 200124 (Other: VUMC IRB)
Record Dates: First submitted 2022-07-28; First posted 2022-08-05 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Autonomic Failure; Pure Autonomic Failure; Multiple System Atrophy; Parkinson Disease; Supine Hypertension; Neurogenic Orthostatic Hypotension
Keywords: CPAP; Hypertension; Orthostatic hypotension
MeSH Terms: conditions — Pure Autonomic Failure; Multiple System Atrophy; Parkinson Disease; Hypertension; Hypotension, Orthostatic | interventions — Sleep; Patient Positioning

STUDY DESIGN:
Intervention Model Description: Randomized, single-blind, crossover
Who Masked: Participant
Masking Description: A sham CPAP will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (5):
- Active CPAP (Daytime Study) (Experimental): CPAP at 8, 10, or 12 cm H2O is applied for up to 2 hours while supine and awake.
  Interventions: Device: Active CPAP
- Sham CPAP (Daytime Study) (Sham Comparator): Sham CPAP is applied for up to 2 hours while supine and awake.
  Interventions: Device: Sham CPAP
- Active CPAP (Overnight Study) (Experimental): CPAP at 8, 10, or 12 cm H2O is applied for up to 9 hours during the night.
  Interventions: Device: Active CPAP
- Sham CPAP (Overnight Study) (Sham Comparator): Sham CPAP is applied for up to 9 hours during the night.
  Interventions: Device: Sham CPAP
- Sleeping in a head-up tilt position (Overnight Study) (Active Comparator): Sleeping with the bed tilted head-up by 10 degrees for up to 9 hours during the night.
  Interventions: Other: Sleeping in a head-up tilt (HUT) position

INTERVENTIONS:
Device: Active CPAP — Continuous positive airway pressure (CPAP) is applied at 8, 10, or 12 cm H20. The active CPAP level will be determined during a CPAP titration trial
  Other Names: Active continuous positive airway pressure
  Arms: Active CPAP (Daytime Study); Active CPAP (Overnight Study)
Device: Sham CPAP — Sham continuous positive airway pressure applied at <4 cm H2O
  Other Names: Sham continuous positive airway pressure
  Arms: Sham CPAP (Daytime Study); Sham CPAP (Overnight Study)
Other: Sleeping in a head-up tilt (HUT) position — Sleeping with the whole bed tilted head-up by 10 degrees or with the head elevated by 13-14 inches.
  Other Names: HUT sleeping
  Arms: Sleeping in a head-up tilt position (Overnight Study)

SUMMARY:
This study aims to learn about the effects of continuous positive airway pressure (CPAP) on people with autonomic failure and high blood pressure when lying down (supine hypertension) to determine if it can be used to treat their high blood pressure during the night. CPAP (a widely used treatment for sleep apnea) involves using a machine that blows air into a tube connected to a mask covering the nose, or nose and mouth, to apply a low air pressure in the airways.

The study includes 3-5 days spent in the Vanderbilt Clinical Research Center (CRC): at least one day of screening tests, followed by up to 3 study days. Subjects may be able to participate in daytime and/or overnight studies. The Daytime study consists of 2 study days: one with active CPAP and one with sham CPAP applied for up to 2 hours. The Overnight study consists of 3 study nights: one with active CPAP, one with sham CPAP, both applied for up to 9 hours and one night sleeping with the bed tilted head-up.

DETAILED DESCRIPTION:
The study includes up to 5 days spent in the Vanderbilt University Medical Center, at least one day of screening tests, followed by 2 study days and/or 2 study nights.

Screening tests include a physical examination and history, routine safety laboratory assessments, and autonomic nervous system testing. Medications for high blood pressure will be held for at least 5 half-lives before studies. Subjects may be able to participate in the daytime and/or the overnight studies.

Daytime Study:

Eligible participants will be studied on two separate days in random order: one day with a high CPAP level and one day with a low CPAP level. The active CPAP level will be determined during a CPAP titration trial

On each study day, participants will be instrumented to measure blood pressure, heart rate, hemodynamic parameters, segmental impedance, and markers of cardiovascular risk. A saline lock or IV catheter will be inserted in one of the arm's veins for blood sample collection. Urine will also be collected during studies.

After baseline measurements, active or sham CPAP will then be applied for up to 2 hours. Outcome measurements will be repeated after 1 and 2 hours of CPAP.

Overnight Studies:

Eligible participants will be studied on three separate nights in random order with a active CPAP, sham CPAP, and sleeping in a head-up tilt position. The active CPAP level will be determined during a CPAP titration trial.

On each study night, the intervention (active CPAP, sham CPAP, or head-up tilt position) will be applied for up to 9 hours. Blood pressure, heart rate, hemodynamic parameters, and markers of cardiovascular risk will be assessed throughout the night. Urine will also be collected during this period. On the following morning, participants will have a tilt table test.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, age 40-80 years, with autonomic failure including pure autonomic failure, multiple system atrophy and Parkinson disease.
* Neurogenic orthostatic hypotension, defined as a ≥20-mmHg decrease in systolic blood pressure within 3 minutes of standing associated with impaired autonomic reflexes determined by autonomic testing in the absence of other identifiable causes.
* Nocturnal supine hypertension (nighttime systolic blood pressure ≥140 mmHg) during the overnight screening for supine hypertension.
* Patients who are willing and able to provide informed consent

Exclusion Criteria:

* Patients with history of recent facial trauma or surgery or intolerance to CPAP or to the CPAP mask.
* Patients who cannot tolerate the medication withdrawal, defined as those who are unable to stand for at least one minute or those with sustained supine blood pressure ≥180/110 mmHg after the medication withdrawal period.
* Bedridden patients or those who are unable to stand due to motor impairment or severe orthostatic hypotension.
* Smokers, patients who are pregnant, or have clinically unstable coronary artery disease, or major cardiovascular or neurological event in the past 6 months; heart failure; and other factors which in the investigator's opinion would prevent the subject from completing the protocol including clinically significant abnormalities in clinical or laboratory testing.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure (daytime) | day 1 and 2 (within 2 hours of the intervention)
  Change from baseline in systolic blood pressure at 2 hours of the intervention
Systolic blood pressure (overnight) | up to 9 hours during the intervention
  Area under the curve of the change from baseline in systolic blood pressure

SECONDARY OUTCOMES:
Stroke Volume (daytime) | day 1 and 2 (within 2 hours of the intervention)
  Change from baseline in stroke volume at 1and 2 hours of the intervention
Natriuretic hormone (daytime) | day 1 and 2 (within 2 hours of the intervention)
  Percent change from baseline in N-terminal-proatrial natriuretic peptide at 2 hours after the intervention
Nocturnal diuresis (overnight) | up to 9 hours during the intervention
  Urine volume collected during the night
Morning orthostatic tolerance (overnight) | during 10 minutes upright tilt
  Area under the curve of the upright systolic blood pressure during head-up tilt

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Autonomic Dysfunction Center/ Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No